CLINICAL TRIAL: NCT04867707
Title: Role of Neuraminidase Activity on Endothelial Dysfunction in Type 2 Diabetes
Acronym: NAED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Luis Martinez-Lemus, DVM, PhD, Professor in Medical Pharmacology Physiology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2038203
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: endothelial dysfunction; vascular function; glycocalyx integrity assessment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Zanamivir

STUDY DESIGN:
Intervention Model Description: Single group design with 20 subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zanamivir treatment (Experimental): Study participants will receive 5 days of treatment with a zanamivir inhaler.
  Interventions: Drug: Zanamivir

INTERVENTIONS:
Drug: Zanamivir — 5 days of treatment with 10mg zanamivir inhaler BID
  Other Names: Relenza

SUMMARY:
The objective is to determine if neuraminidase inhibition with zanamivir is efficacious as a therapeutic strategy to restore endothelial function in T2D patients.

DETAILED DESCRIPTION:
Twenty subjects will complete five days of treatment with zanamivir. Baseline measurements will be taken before the initiation of treatment, as well as after the conclusion of the treatment period (i.e., a total of two assessment visits per subject). Assessment visits will include: vitals (such as blood pressure, heart rate), fasting blood work for plasma neuraminidase activity, plasma sialic acid, plasma glucose and plasma insulin, brachial artery FMD, and glycocalyx integrity assessment via Glycocheck.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with a BMI of 25-39 kg/m2
2. Ages 45-64 years at randomization.
3. Diagnosis of T2D classified based on physician diagnosis.
4. No vulnerable populations (e.g., prisoners, pregnant, children) will be enrolled.

Exclusion Criteria:

1. Cardiovascular disease including myocardial infraction, heart failure, coronary artery disease, stroke
2. History of chronic renal or hepatic disease
3. Active cancer
4. Autoimmune diseases
5. Immunosuppressant therapy
6. Hormone replacement therapy
7. Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
8. Current tobacco use
9. Pregnancy (Premenopausal women will be required to complete a urine pregnancy test before participation)
10. History of asthma or chronic obstructive pulmonary disease.
11. History of allergic reaction to lactose or milk proteins
12. Intranasal live attenuated influenza vaccine (LAIV) given within 2 weeks before zanamivir administration or a planned dose within 48 hours after zanamivir administration. Product insert states to avoid zanamivir administration with intranasal live attenuated influenza vaccine (LAIV).

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Martinez-Lemus, PhD, Principal Investigator — University of Missouri, School of Medicine
Locations (1):
- University of Missouri, School of Medicine Clinical Research Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foote CA, Ramirez-Perez FI, Smith JA, Ghiarone T, Morales-Quinones M, McMillan NJ, Augenreich MA, Power G, Burr K, Aroor AR, Bender SB, Manrique-Acevedo C, Padilla J, Martinez-Lemus LA. Neuraminidase inhibition improves endothelial function in diabetic mice. Am J Physiol Heart Circ Physiol. 2023 Dec 1;325(6):H1337-H1353. doi: 10.1152/ajpheart.00337.2023. Epub 2023 Oct 6. PMID 37801046

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zanamivir Treatment
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zanamivir Treatment
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycocalyx Integrity-Perfused Boundary Region
Description: Glycocalyx integrity will be assessed non-invasively using the GlycoCheck. The Glycocheck video microscope instrument will be placed under the subject's tongue to assess red blood cell penetration of the glycocalyx lining. PBR (perfused boundary region) is a measure of distance (mcm) that red blood cells penetrate into the glycocalyx. An increase in PBR in indicative of lower glycocalyx integrity. Outcomes are reported as a change in PBR from Day 0 to Day 5.
Time Frame: Day 0 and Day 5
Population: participants that completed full study intervention with baseline and day 5 assessment.
Measure: Mean (Standard Error); unit: micrometers (mcm)
Arm/Group | Zanamivir Treatment
Number analyzed (Participants) | 14
micrometers (mcm) | -0.0057 (0.11)

ADVERSE EVENTS:
Time Frame: Baseline assessment (day 0) through Final assessment (Day 5)
Description: Participants were administered a side effects and toxicity questionnaire daily during the dosing period. The questionnaire assessed for common side effects of zanamivir listed in the packaging insert.
Arm/Group | Zanamivir Treatment
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanamivir Treatment (N=14)
Changes in mood, sleep, or appetite (General disorders) | 4 (6)
Sinus congestion and inflammation (General disorders) | 0 (0)
Coughing, tightness in chest, wheezing, SOB, difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Joint pain/swelling (Musculoskeletal and connective tissue disorders) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0)
Dizziness (General disorders) | 0 (0)
Fever/Chills (General disorders) | 0 (0)
Hallucinations or delusions (Psychiatric disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT04867707/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04867707/ICF_001.pdf